CLINICAL TRIAL: NCT02600702
Title: A Randomized Control Study of Siriraj Home Exercises Protocol for Primary Knee Osteoarthritis Patients Versus Usual Orthopedic Outpatient Consultation in Primary Knee Osteoarthritis Patients
Brief Title: A Study of Siriraj Home Exercises Protocol for Primary Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 444/2557(EC4)
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Home base exercise
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- usual care (No Intervention): quadricep exercise
- Siriraj home base exercise (Experimental): Knee exercise protocol for 12 position for 3 months with low-impact aerobic exercise
  Interventions: Other: Siriraj knee exercise
- Modalities and exercise (Active Comparator): Physical modalities for 6 weeks and Knee exercise protocol for 12 position for 3 months with low-impact aerobic exercise
  Interventions: Other: Siriraj knee exercise; Other: Physical modalities

INTERVENTIONS:
Other: Siriraj knee exercise — Siriraj knee exercise, 12 position of exercise protocol
  Arms: Modalities and exercise; Siriraj home base exercise
Other: Physical modalities
  Arms: Modalities and exercise

SUMMARY:
The purpose of this study is to compare the exercise protocol called "Siriraj home base exercise program for OA knee" to usual care and physical modalities for conservative treatment in patients with 1st OA knee.

ELIGIBILITY:
Inclusion Criteria:

* 1st osteoarthritis of the knee Age >/= 50 yrs

Exclusion Criteria:

* Previous knee surgery for OA knee treatment
* Has plan or schedule for knee surgery
* Severe degree of OA knee.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
WOMAC score | 3 months

SECONDARY OUTCOMES:
6 mins walk test | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj hospital, Bangkok, Thailand